CLINICAL TRIAL: NCT06584747
Title: Study of Cerebral Vascular Reserve Using Pharmacological Testing With Acetazolamide: A Non-Inferiority Study of PET Method Compared to Conventional Reference Scintigraphy
Acronym: DIAMOX-TEP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024/27
Record Dates: First submitted 2024-08-27; First posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Cerebrovascular Circulation
MeSH Terms: interventions — Positron-Emission Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental Arms (Experimental)
  Interventions: Diagnostic Test: PET scan

INTERVENTIONS:
Diagnostic Test: PET scan — 18F-FDG PET scans will be performed to assess cerebral vascular reserve. For exams involving stimulation with Acetazolamide (DIAMOX®), the radiopharmaceutical injection (18F-FDG or 99mTc-HMPAO) will start exactly 15 minutes after the Acetazolamide (DIAMOX®) injection.

SUMMARY:
This study compares two methods for assessing brain blood flow. PET scan will be use with a drug called Acetazolamide and compare its effectiveness to the standard scintigraphy method. The goal is to see if the PET scan is just as good as the traditional method in measuring how well the brain's blood vessels respond to the drug.

ELIGIBILITY:
Inclusion Criteria:

* Chronic stenosing cerebral vascular pathology (stenosis > 70% on Doppler examination or angiography).
* Patient aged over 18 years.
* Patient who has voluntarily agreed to participate in the study and has signed the written informed consent.
* Patient affiliated with a social security system.

Exclusion Criteria:

* Patient with stenosis less than 70% on Doppler examination or angiography.
* Patient with a contraindication to 18F-FDG PET examinations: severe claustrophobia, poorly controlled diabetes during 18F-FDG PET examinations (fasting capillary blood glucose ≥ 11 mmol/L).
* Patient with a contraindication to scintigraphy.
* Patient with an allergy to sulfonamides (Acetazolamide DIAMOX®).
* Patient enrolled in another clinical study with a specified exclusion period.
* Minor patient.
* Patient unable to give informed consent.
* Vulnerable individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
diagnostic performance of the 18F-FDG PET | 12 months
  The primary endpoint is the sensitivity of the examination in detecting a decrease in cerebral vascular reserve (CVR). The presence or absence of a decrease in CVR for each patient will be determined by clinical consensus, based in particular on spontaneous follow-up (clinical progression, cerebral ischemic episodes, etc.) and/or on the progression after revascularization in cases where it is performed.

SECONDARY OUTCOMES:
contribution of late 18F-FDG PET metabolic information | 12 months
  To study the contribution of late 18F-FDG PET metabolic information: Late 18F-FDG PET metabolic images will be analyzed using Scenium® software, which enables stereotaxic normalization and the expression of uptake in terms of standard deviations relative to a database of normal subjects. The corresponding values will be compared based on the clinical progression of patients after revascularization.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Antoine Lacassagne, Nice, France

IPD SHARING:
Plan to Share IPD: Undecided